CLINICAL TRIAL: NCT06104358
Title: A 6-Month, Randomized, Double-Blind, Placebo-controlled, Phase 2a Study of the Effects of HU6 on Energy Metabolism, Muscle and Liver Substrate Metabolism, and Mitochondrial Function in Subjects Who Are Overweight or Obese With Type 2 Diabetes
Brief Title: Ph 2a Study of HU6 on Energy Metabolism, Muscle and Liver Substrate Metabolism, and Mitochondrial Function in Subjects Who Are Overweight or Obese With Type 2 Diabetes
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The protocol was redirected by the FDA to another division and will be resubmitted at a future date.
Sponsor: Rivus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RIV-HU6-204
Record Dates: First submitted 2023-10-11; First posted 2023-10-27 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Diabete Type 2; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active Treatment HU6 (Experimental): Subjects who are randomized to active study drug will receive 450mg of HU6 for 14 day and then 600mg of HU6 for 168 days. N = 24
  Interventions: Drug: HU6
- Placebo (Placebo Comparator): Placebo Comparator is non-active study drug. N = 24
  Interventions: Drug: HU6

INTERVENTIONS:
Drug: HU6 — HU6 is being evaluated for its effect on Energy Metabolism, Muscle and Liver Substrate Metabolism, and Mitochondrial Function

SUMMARY:
This is a randomized, double-blind, placebo-controlled parallel group study of HU6 and placebo in subjects who are overweight or obese with T2D.

The study will be conducted in 4 stages.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled parallel group study of HU6 and placebo in subjects who are overweight or obese with T2D.

The study will be conducted in 4 stages (Figure 1).

* Stage 1: (screening) is conducted over a 29-day window (Day -48 to Day -20). Subjects who meet all of the eligibility criteria may proceed Stages 2 to 4 of the study.
* Stage 2 (baseline [pre-randomization]) is conducted over a 19-day period prior to randomization and includes a 13-day run-in and the first 6-day inpatient assessment period. At the end of Stage 2, subjects will be randomized 1:1 to HU6 or placebo.
* Stage 3 (double-blind dosing) is conducted after randomization. Day 1 is the first dose of double-blind study drug, and dosing continues over an approximate 26-week period. During this time, there will be study visits for safety, PK, and PD. Stage 3 of the study concludes with a 3-day run-in followed by the second 6-day inpatient assessment period.
* Stage 4 (washout) is conducted after dosing has ended and includes an approximate 4-week washout duration including a 3-day run-in followed by the third inpatient assessment period (3-day duration). The last day of the 3-day inpatient stay is the end-of-study. (Note that there will be a separate early termination visit for any subject who prematurely discontinues from the study

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand the procedures and requirements of the study and provide written informed consent and authorization for protected health information disclosure.
2. Willing and able to comply with the requirements of the study protocol.
3. Male or female 18 to 70 years of age, inclusive, at time of informed consent.
4. Body mass index (BMI) >28.0 kg/m2 and able to fit into the MRI machine.
5. Subject has T2D meeting all of the following criteria:

Exclusion Criteria:

1. Body weight >450 pounds.
2. Subject-reported history of weight gain or loss >5% in 3 months prior to screening.
3. The subject participates in programmed exercise >3 hours per week.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-11-17 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Sleeping Metabolic Rate (SMR) change from Baseline to 6 Months (26 weeks) | 26 weeks
  Change from baseline in SMR at 6 months (26 weeks) as assessed by whole room indirect calorimetry (WRIC).

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Garner, PhD, Study Director — Rivus Pharmaceuticals, Inc.
Locations (1):
- AdventHealth Translational Research Institute, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided